CLINICAL TRIAL: NCT01681433
Title: The Pacific Clinical Trial: A Randomized Phase II Study Evaluating OGX-427 in Patients With Metastatic Castrate-Resistant Prostate Cancer (MCRPC)Who Have Prostate-Specific Antigen (PSA) Progression While Receiving Abiraterone: Hoosier Oncology Group GU12-159
Brief Title: OGX-427 in Metastatic Castrate-Resistant Prostate Cancer With Prostate-Specific Antigen Progression While Receiving Abiraterone
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: Costantine Albany (Other)
Collaborators: Hoosier Cancer Research Network (Other); Achieve Life Sciences (Industry)
Responsible Party: Sponsor-Investigator, Costantine Albany, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GU12-159
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer; Metastatic Castrate-Resistant Prostate Cancer; PSA
Keywords: OGX-427; Abiraterone Acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apatorsen; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Arm A (Experimental): OGX-427 + continuation of standard therapy with abiraterone acetate and prednisone
  Interventions: Drug: OGX-427; Drug: Abiraterone Acetate; Drug: Prednisone
- Control Arm: Arm B (Active Comparator): Continuation of standard therapy with abiraterone acetate and prednisone
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone

INTERVENTIONS:
Drug: OGX-427 — OGX-427 started within 7 days of randomization, three loading doses of 600 mg IV within Week 1 if possible (up to 10 days of initiating treatment), followed by weekly doses of 800 mg IV
  Arms: Experimental: Arm A
Drug: Abiraterone Acetate — Standard therapy: Abiraterone Acetate 1000 mg PO daily
Drug: Prednisone — Standard therapy: Prednisone 10-20 mg PO daily

SUMMARY:
This Phase II study has been designed to evaluate the anti-tumor effects of adding OGX-427 to continuing abiraterone acetate and prednisone treatment in men with metastatic castrate-resistant prostate cancer (MCRPC) who have prostate-specific antigen (PSA) progression

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

This is an open-label, randomized, Phase II clinical trial designed to evaluate the anti-tumor effects of OGX-427 and continuing abiraterone acetate and prednisone versus continuing abiraterone acetate and prednisone alone in men with MCRPC who have evidence of PSA progression but no evidence of symptomatic or radiographic progression that would require alternative therapy (e.g., needing radiation therapy for pain or significant progression of visceral metastases).

Patients on the control arm will be allowed to cross-over to receive OGX-427 following documented disease progression. Patients will be randomized with equal probability to one of the following arms:

EXPERIMENTAL ARM (Arm A):

OGX-427 Starting within 7 days of randomization, three loading doses of 600 mg intravenously (IV) within Week 1 if possible (up to 10 days of initiating treatment), followed by weekly doses of 800 mg IV

Continuation of standard therapy with abiraterone acetate 1000 mg by mouth (PO) daily and prednisone 10-20 mg PO daily

CONTROL ARM (Arm B):

Continuation of standard therapy with abiraterone acetate 1000 mg PO daily and prednisone 10-20 mg PO daily

After documented disease progression, patients on Arm B may opt to receive OGX-427 treatment (according to the Arm A schedule) following a screening evaluation (i.e., all inclusion and exclusion criteria have been met)

Both Arms:

Evaluations at 4 week-intervals. Disease assessments required at the milestone Day 60 assessment (expected to occur after 8 weeks of treatment and prior to Day 1, Week 9) and at 16, 24, 32, 40, and 48 weeks (if applicable) or until documented disease progression. Patients who are withdrawn from the study for a reason other than documented disease progression or patient withdrawal of consent will be followed every 4 weeks in the Off-Treatment Follow-up Period until documented disease progression.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Life Expectancy: Not Specified

Hematopoietic:

* Absolute neutrophil count (ANC) ≥ 1.5 x 109 cells /L, platelet count ≥ 100 x 109 /L, and hemoglobin ≥ 9 g/dL without transfusion

Hepatic:

* Total bilirubin ≤ 1.1 x upper limit of normal (ULN) unless elevated secondary to conditions such as Gilbert's disease, in which case a direct bilirubin ≤ ULN is required
* Serum glutamic pyruvic transaminase (SGPT), alanine transaminase (ALT) and alanine transaminase (SGOT) aspartate transaminase (AST) ≤ 3.0 x ULN

Renal:

* Creatinine ≤ 1.3 x ULN

Cardiac:

* Known left ventricular ejection fraction (LVEF) <50% or New York Heart Association (NYHA) Functional Classification Class III or IV heart failure

Other:

* Castrate serum testosterone level (< 50 ng/dL or < 1.7 nmol/L)
* Potassium within normal limits

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the following criteria to be eligible for inclusion into the study.

* Histological or cytological diagnosis of adenocarcinoma of the prostate
* Metastatic disease on chest, abdominal, or pelvic computed tomography (CT) scan and/or bone scan
* Currently receiving abiraterone acetate and prednisone and meeting the following criteria:

  * Any PSA decline within 12 weeks from initiation of abiraterone acetate
  * Currently tolerating abiraterone acetate (1000 mg oral daily) and prednisone (10-20 mg oral daily)
  * PSA progression, defined as an increase in PSA which is ≥25% above the nadir and an absolute value of ≥2 ng/mL, which is confirmed by a second value ≥2 weeks later.
  * No evidence of symptomatic or radiographic progression that would require alternative therapy (e.g., needing radiation therapy for pain or significant progression of visceral metastases or >33% increase in daily opioid use within 2 weeks prior to randomization).
* All patients who have not had a surgical orchiectomy must continue treatment with a luteinizing hormone-releasing hormone (LHRH) agonist or antagonist to maintain a castrate level of testosterone.
* Patient must fulfill "Prior Therapy" criteria as follows:

  * Chemotherapy: no more than 1 prior chemotherapy regimen for castrate-resistant prostate cancer (CRPC) is permitted; a minimum of at least 28 days must have passed since the last dose of chemotherapy.
  * Hormone therapy: hormonal androgen ablation therapy prior to abiraterone is required.
  * Experimental therapy: prior non-cytotoxic experimental therapy is permitted provided a minimum of at least 14 days has passed since completing therapy. Prior treatment with enzalutamide (MDV3100) is allowed.
  * Radiation: prior external beam radiation is permitted provided a minimum of at least 14 days have passed since completing radiotherapy (exception for radiotherapy: at least 7 days since completing a single fraction of ≤800 cGy to a restricted field or limited-field radiotherapy to non-marrow bearing area such as an extremity or orbit) at the time of randomization
* Must be willing to use effective contraception throughout study treatment and for 3 months after completion of study treatment if able to father a child.
* Must be willing not to change (add or subtract) bone protecting therapy (bisphosphonates and/or denosumab) during the study unless changed for toxicity.
* Written informed consent must be obtained prior to any protocol-specific procedures being performed.

Exclusion Criteria:

Subjects meeting ANY of the following exclusion criteria will NOT be eligible for inclusion into the study:

* Currently receiving abiraterone acetate in combination with any other anti-cancer agent (except prednisone)
* Documented brain metastases, or carcinomatous meningitis, treated or untreated (Brain imaging for asymptomatic patients is not required.)
* Cord compression requiring surgery or radiation therapy while on abiraterone treatment
* Active second malignancy (including lymphoid malignancies such as chronic lymphocytic leukemia or low grade lymphoma) defined, in general, as requiring anticancer therapy or at high risk of recurrence during the study; not including adequately treated non melanomatous skin cancer or other solid tumors curatively treated with no evidence of disease in > 3 years
* History of allergic reactions to therapeutic antisense oligonucleotides
* Active autoimmune disease requiring treatment
* Participated in a prior Phase 3 clinical study evaluating custirsen regardless of study arm assignment (i.e., either control or investigational arm), or prior exposure to OGX-427
* Uncontrolled medical conditions such as myocardial infarction, uncontrolled hypertension, stroke or treatment of a major active infection within 3 months of randomization, as well as any significant concurrent medical illness that in the opinion of the Investigator would preclude protocol therapy
* Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device. Concomitant participation in observational studies is acceptable.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Albany, M.D., Principal Investigator — Hoosier Cancer Research Network
Locations (16):
- United States (10):
  - Prostate Oncology Specialists, Inc., Marina del Rey, California
  - IU Health Bloomington Hospital, Bloomington, Indiana
  - IU Health Goshen Hospital, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of New Mexico Cancer Center: Albuquerque, Albuquerque, New Mexico
  - Virginia Oncology Associates, Norfolk, Virginia
- Canada (6):
  - Alberta Health Services: Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim N. Chi, Christopher Sweeney, Cindy Jacobs, Patricia S. Stewart, Noah M. Hahn. The Pacific trial: A randomized phase II study of OGX-427 in men with metastatic castration-resistant prostate cancer (mCRPC) and PSA progression while receiving abiraterone acetate (AA). J Clin Oncol 31, 2013 (suppl; abstr TPS5101) http://abstracts2.asco.org/AbstView_132_115104.html
- See also: Hoosier Cancer Research Network Website — https://hoosiercancer.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: Arm A | Control Arm: Arm B
Started | 36 | 36
Completed | 4 | 3
Not Completed | 32 | 33
Not completed — Lack of Efficacy | 23 | 23
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Protocol Violation | 2 | 0
Not completed — Adverse Event | 2 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Arm A | Control Arm: Arm B | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Median (Full Range); unit: years] | 71 [53 to 85] | 72 [57 to 89] | 72 [53 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 36 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 30 | 28 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 14 | 15 | 29
  United States | 22 | 21 | 43
ECOG Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  participants
    ECOG 0 | 16 | 16 | 32
    ECOG 1 | 20 | 20 | 40
Median PSA [Median (Full Range); unit: ug/L] | 34.19 [2.51 to 387.60] | 18.17 [4.24 to 302.15] | 23 [2.51 to 387.60]

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: To ascertain whether Arm A has a greater proportion of patients observed to be alive without progression at Day 60 (±7 days) as compared to Arm B.
Time Frame: 60 days
Measure: Number; unit: participants
Arm/Group | Experimental: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 36 | 36
participants | 12 | 6

2. Secondary Outcome: PSA Response
Description: Compare arms to determine the proportion of patients who have a PSA response (≥ 30% decline) and any PSA decline post-randomization.
Time Frame: 60 days
Measure: Number; unit: participants
Arm/Group | Experimental: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 36 | 36
participants
  PSA DECLINE >= 30% | 2 | 2
  PSA DELCINE >=50 % | 2 | 1
  ANY DECLINE | 13 | 11

3. Other Pre Specified Outcome: Objective Response
Description: Compare arms to determine the objective response of study patients, per RECIST 1.1
Time Frame: 60 days
Measure: Number; unit: participants
Arm/Group | Experimental: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 33 | 30
participants
  Partial Response | 1 | 0
  Stable Disease | 6 | 5
  Progressive Disease | 26 | 25

4. Other Pre Specified Outcome: Time to Disease Progression
Description: Compare arms to determine the time to disease progression of study patients
Time Frame: 60 days
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 36 | 36
months | 1.9055 [1.0842 to 2.32341] | 1.0842 [.9856 to 1.8398]

5. Other Pre Specified Outcome: Circulating Tumor Cell (CTC) Counts
Description: Compare arms to determine circulating tumor cell (CTC) counts for patients at baseline and while on study
Time Frame: Every 4 weeks
Measure: Number; unit: participants
Arm/Group | Experimental: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 32 | 30
participants
  Best CTC Change from Baseline >=5 to <5 | 8 | 4
  Best CTC Change from Baseline <5 to <5 | 16 | 15
  Best CTC Change from Baseline >=5 to >=5 | 7 | 10
  Best CTC Change from Baseline<5 to >=5 | 1 | 1

6. Other Pre Specified Outcome: Protein Levels
Description: Compare arms to determine levels of heat shock protein 27 (Hsp27), clusterin, and other relevant proteins of patients at baseline and during study
Time Frame: Every 4 weeks
Population: Data for this secondary objective was not collected or analyzed
Arm/Group | Experimental: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Phosphatase and Tensin Homolog (PTEN) Deletion Status
Description: Compare arms to determine PTEN deletion status in original pathology specimens correlated with clinical outcomes
Time Frame: Every 4 weeks
Population: Data for this objective was not collected or analyzed
Arm/Group | Experimental: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Every four weeks, up to 48 weeks or disease progression.
Description: All adverse events for all subjects who were both randomized to arm A and crossed over to Arm A. 20 subjects crossed over to arm A after disease progression and their adverse events are reported from the date of crossover.
Arm/Group | Experimental: Arm A | Control Arm: Arm B
All-Cause Mortality (participants affected / at risk) | 8/56 | 6/36
Serious Adverse Events (participants affected / at risk) | 12/56 | 6/36
Other Adverse Events (participants affected / at risk) | 51/56 | 32/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Arm A (N=56) | Control Arm: Arm B (N=36)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0)
CONFUSION (Psychiatric disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EDEMA LIMBS (General disorders) | 1 (1) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 2 (2) | 0 (0)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 3 (3) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 1 (1) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 2 (2) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (3) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Arm A (N=56) | Control Arm: Arm B (N=36)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 2 (2)
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 1 (1)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 9 (17) | 0 (0)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (7) | 1 (1)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 13 (25) | 10 (12)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 5 (6) | 9 (15)
ANXIETY (Psychiatric disorders) | 4 (4) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 8 (18) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 15 (21) | 12 (15)
BLADDER INFECTION (Infections and infestations) | 2 (3) | 0 (0)
BLADDER SPASM (Renal and urinary disorders) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 6 (11) | 6 (7)
BRONCHIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BRUISING (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
CHILLS (General disorders) | 16 (23) | 3 (4)
CHOLESTEROL HIGH (Investigations) | 4 (4) | 7 (7)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1) | 0 (0)
CONFUSION (Psychiatric disorders) | 1 (2) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 6 (6) | 10 (12)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 10 (12)
CREATININE INCREASED (Investigations) | 3 (5) | 1 (1)
CUSHINGOID (Endocrine disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
DEPRESSION (Psychiatric disorders) | 3 (3) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 11 (14) | 8 (14)
DIZZINESS (Nervous system disorders) | 7 (7) | 1 (2)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 2 (2)
DYSPHASIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 8 (20) | 6 (9)
EDEMA LIMBS (General disorders) | 8 (9) | 7 (8)
EDEMA TRUNK (General disorders) | 1 (1) | 2 (3)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
EXTERNAL EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0)
EYE DISORDERS (Eye disorders) | 2 (2) | 2 (2)
FACIAL PAIN (General disorders) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
FATIGUE (General disorders) | 26 (40) | 22 (32)
FEVER (General disorders) | 11 (12) | 2 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
FLU LIKE SYMPTOMS (General disorders) | 4 (4) | 1 (1)
FLUSHING (Vascular disorders) | 3 (3) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 2 (2)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 1 (1) | 2 (4)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 8 (10) | 3 (4)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (6) | 6 (7)
GLAUCOMA (Eye disorders) | 2 (2) | 1 (1)
HEADACHE (Nervous system disorders) | 8 (9) | 5 (5)
HEMATURIA (Renal and urinary disorders) | 1 (1) | 3 (3)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 2 (2)
HEPATITIS VIRAL (Infections and infestations) | 2 (2) | 0 (0)
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 1 (1) | 1 (1)
HOT FLASHES (Vascular disorders) | 3 (3) | 4 (5)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 (6) | 5 (8)
HYPERTENSION (Vascular disorders) | 12 (17) | 18 (19)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
HYPOKALEMIA (Metabolism and nutrition disorders) | 11 (16) | 5 (13)
HYPONATREMIA (Metabolism and nutrition disorders) | 3 (4) | 2 (4)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
HYPOTENSION (Vascular disorders) | 4 (5) | 2 (2)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 2 (2)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 2 (2) | 2 (2)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 6 (7)
INVESTIGATIONS (Investigations) | 1 (1) | 0 (0)
LARYNGEAL HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LOCALIZED EDEMA (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0)
MUCOSITIS ORAL (Gastrointestinal disorders) | 2 (2) | 0 (0)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 25 (28) | 9 (11)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 3 (4) | 2 (3)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (8) | 1 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (3) | 1 (1)
PAIN (General disorders) | 7 (8) | 10 (12)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 (9) | 14 (21)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1) | 0 (0)
PARESTHESIA (Nervous system disorders) | 1 (1) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 (3) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 6 (6) | 7 (9)
PLATELET COUNT DECREASED (Investigations) | 5 (11) | 3 (6)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PURPURA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 5 (5) | 2 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
RESTLESSNESS (Psychiatric disorders) | 2 (2) | 0 (0)
SINUSITIS (Infections and infestations) | 2 (3) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SPASTICITY (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 1 (1)
URINARY FREQUENCY (Renal and urinary disorders) | 2 (2) | 8 (9)
URINARY INCONTINENCE (Renal and urinary disorders) | 2 (3) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 6 (6)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2)
URINARY TRACT PAIN (Renal and urinary disorders) | 2 (2) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
URINE OUTPUT DECREASED (Investigations) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR DISORDERS (Vascular disorders) | 1 (1) | 2 (2)
VASOVAGAL REACTION (Nervous system disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 2 (2) | 0 (0)
VITREOUS HEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 15 (18) | 7 (8)
WEIGHT LOSS (Investigations) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 2 (6)
CARDIAC DISORDERS (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC TROPONIN I INCREASED (Investigations) | 0 (0) | 1 (1)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 0 (0) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENDOCRINE DISORDERS (Endocrine disorders) | 0 (0) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 2 (2)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GYNECOMASTIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
HEARING IMPAIRED (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HYPERPARATHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ILEAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
LIBIDO DECREASED (Psychiatric disorders) | 0 (0) | 3 (3)
LYMPHOCYTE COUNT INCREASED (Investigations) | 0 (0) | 1 (1)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NIGHT BLINDNESS (Eye disorders) | 0 (0) | 1 (1)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PROCTITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
RENAL CALCULI (Renal and urinary disorders) | 0 (0) | 1 (1)
RETINAL VASCULAR DISORDER (Eye disorders) | 0 (0) | 1 (1)
RHINITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1)
SCROTAL PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (2)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
STOMACH PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
SURGICAL AND MEDICAL PROCEDURES (Surgical and medical procedures) | 0 (0) | 1 (1)
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 (0) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
WEIGHT GAIN (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT01681433/Prot_SAP_000.pdf